CLINICAL TRIAL: NCT05025215
Title: Study on the Effect of Precise Aerosol Inhalation Nursing Program on Effective Sputum Excretion in Elderly Patients With Lung Surgery
Brief Title: The Effect of Precise Aerosol Inhalation Nursing on Sputum Excretion in Elderly Patients With Lung Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210822
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A： Precise (Experimental): The experimental group accepts improved precise aerosol inhalation nursing program，which was based on the traditional oxygen aerosol inhalation treatment, including precise body position care, time control, observation and treatment, evaluation, etc. This group is planned to enroll 100 patients.
  Interventions: Behavioral: Precise Aerosol Inhalation Nursing Program
- Group B：Traditional (Experimental): The control group accepts traditional aerosol inhalation nursing method. This group is planned to enroll 100 patients.
  Interventions: Behavioral: Traditional Aerosol Inhalation Nursing Method

INTERVENTIONS:
Behavioral: Precise Aerosol Inhalation Nursing Program — The precise aerosol inhalation nursing program was based on the traditional oxygen aerosol inhalation treatment, including precise body position care, time control, observation and treatment, evaluation, etc.
  Arms: Group A： Precise
Behavioral: Traditional Aerosol Inhalation Nursing Method — The traditional aerosol inhalation nursing method is carried out according to the operation of aerosol inhalation.
  Arms: Group B：Traditional

SUMMARY:
Comparing the effects of different kinds of aerosol inhalation nursing programs on effective sputum excretion in elderly patients with lung surgery.

DETAILED DESCRIPTION:
Based on the traditional oxygen aerosol inhalation treatment, this study will improve it. In the process, precise body position care, time control, observation and treatment, evaluation, etc. will be used to form a precise aerosol inhalation care plan. To explore the effect of this program on effective sputum excretion in elderly patients undergoing lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* ①The patient underwent thoracoscopic lung surgery; ②There was no obvious pulmonary infection before the operation; ③Good audiovisual function, no communication barriers, able to cooperate with nebulized inhalation operation; ④Patients informed consent to this study.

Exclusion Criteria:

* ①Patients with mental illness; ②Acute COPD; ③Serious complications or failure of important organs after operation.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-08 (Actual); Primary Completion 2022-05-08 (Estimated); Study Completion 2022-05-08 (Estimated)

PRIMARY OUTCOMES:
Standardization of aerosol inhalation | From the first to the third day after surgery.
  The investigators use a self-made inhalation implementation standard evaluation form to evaluate whether inhalation was standard in postoperative patients.

SECONDARY OUTCOMES:
Adverse events | From the first to the third day after surgery.
  Discomfort during inhalation: chest tightness, dyspnea, palpitations, elevated blood pressure, etc.
Viscosity of sputum | From the first to the third day after surgery.
  According to the viscosity, the sputum was divided into three types: ⅰ degree (thin phlegm), ⅱ degree (moderate phlegm), ⅲ degree (severe phlegm).
Phlegm retention | From the first to the third day after surgery.
  Sputum sounds can be heard or ausculted at the bedside.
Patient satisfaction | The third day after surgery.
  Likert 5-level scoring method was adopted to allow patients to evaluate the nursing plan. The higher the score, the more satisfied the patients were.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Luo, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosnic-Anticevich SZ, Sinha H, So S, Reddel HK. Metered-dose inhaler technique: the effect of two educational interventions delivered in community pharmacy over time. J Asthma. 2010 Apr;47(3):251-6. doi: 10.3109/02770900903580843. PMID 20394511
- [Background] Press VG, Kelly CA, Kim JJ, White SR, Meltzer DO, Arora VM. Virtual Teach-To-Goal Adaptive Learning of Inhaler Technique for Inpatients with Asthma or COPD. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1032-1039.e1. doi: 10.1016/j.jaip.2016.11.018. Epub 2017 Jan 5. PMID 28065689
- [Background] Pedersen S, Ostergaard PA. Nasal inhalation as a cause of inefficient pulmonal aerosol inhalation technique in children. Allergy. 1983 Apr;38(3):191-4. doi: 10.1111/j.1398-9995.1983.tb01605.x. PMID 6846746
- [Background] Fink JB, Rubin BK. Problems with inhaler use: a call for improved clinician and patient education. Respir Care. 2005 Oct;50(10):1360-74; discussion 1374-5. PMID 16185371
- [Background] Klijn SL, Hiligsmann M, Evers SMAA, Roman-Rodriguez M, van der Molen T, van Boven JFM. Effectiveness and success factors of educational inhaler technique interventions in asthma & COPD patients: a systematic review. NPJ Prim Care Respir Med. 2017 Apr 13;27(1):24. doi: 10.1038/s41533-017-0022-1. PMID 28408742
- [Background] Wu M, Woodrick NM, Arora VM, Farnan JM, Press VG. Developing a Virtual Teach-To-Goal Inhaler Technique Learning Module: A Mixed Methods Approach. J Allergy Clin Immunol Pract. 2017 Nov-Dec;5(6):1728-1736. doi: 10.1016/j.jaip.2017.04.032. Epub 2017 Jun 7. PMID 28600133
- [Background] Price DB, Roman-Rodriguez M, McQueen RB, Bosnic-Anticevich S, Carter V, Gruffydd-Jones K, Haughney J, Henrichsen S, Hutton C, Infantino A, Lavorini F, Law LM, Lisspers K, Papi A, Ryan D, Stallberg B, van der Molen T, Chrystyn H. Inhaler Errors in the CRITIKAL Study: Type, Frequency, and Association with Asthma Outcomes. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1071-1081.e9. doi: 10.1016/j.jaip.2017.01.004. Epub 2017 Mar 9. PMID 28286157
- [Background] Press VG, Arora VM, Trela KC, Adhikari R, Zadravecz FJ, Liao C, Naureckas E, White SR, Meltzer DO, Krishnan JA. Effectiveness of Interventions to Teach Metered-Dose and Diskus Inhaler Techniques. A Randomized Trial. Ann Am Thorac Soc. 2016 Jun;13(6):816-24. doi: 10.1513/AnnalsATS.201509-603OC. PMID 26998961
- [Background] Press VG, Arora VM, Shah LM, Lewis SL, Charbeneau J, Naureckas ET, Krishnan JA. Teaching the use of respiratory inhalers to hospitalized patients with asthma or COPD: a randomized trial. J Gen Intern Med. 2012 Oct;27(10):1317-25. doi: 10.1007/s11606-012-2090-9. Epub 2012 May 17. PMID 22592354